CLINICAL TRIAL: NCT00999999
Title: Fleece Bound Tissue Sealing With TachoSil® to Assist in Closing of the Dura Mater After Elective Craniotomy to Reduce Postoperative Cerebrospinal Fluid (CSF) Leakage.
Brief Title: Efficacy of Tachosil as Dural Sealant Compared to Standard Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Nycomed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Tachousb-1; EKBB 182/09 (Other: EKBB); Swissmedic 2009DR4198 (Other: Swissmedic)
Record Dates: First submitted 2009-10-21; First posted 2009-10-22 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: Subjects Scheduled for Supra-/Infratentorial Craniotomy
Keywords: Craniotomy outcome; CSF leakage; Dural sealant
MeSH Terms: conditions — Cerebrospinal Fluid Rhinorrhea

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard (Active Comparator): Standard dural closure
  Interventions: Procedure: Craniotomy supra- or infratentorial, dural closure
- Experimental (Experimental): Experimental dural closure, adding of Investigational Medicinal Product (IMP)
  Interventions: Procedure: Craniotomy supra- or infratentorial, dural closure

INTERVENTIONS:
Procedure: Craniotomy supra- or infratentorial, dural closure — After dural closure with a water-tight suture, randomization is performed. Depending on the randomization outcome, the study drug Tachosil is applied on the dural suture or omitted.

SUMMARY:
Main objective of this trial is to assess the hypothesis whether the application of TachoSil® as a dural sealant improves the quality of craniotomy procedure and outcome in general compared with standard dural closure techniques in a controlled and randomized way. As a primary endpoint the investigators look at possible postoperative occurrence of CSF pads or leakages needing any kind of intervention until day 30 after the primary craniotomy. Furthermore, the investigators will look at other surgery-related complications and at pharmacoeconomic endpoints such as hospital stay or cost of the implant. Overall, the results of this study will provide important information on whether or not the adjunct of a relatively expensive implant on a routinely basis for the closure of elective craniotomies is safe and effective, or not.

To date, TachoSil® is often used in neurosurgery and other surgical disciplines in a non-standardized fashion also to prevent CSF leakage after dural closure. So far, adverse events directly related to the product have not been reported. Theoretically, any implant may be associated with a higher incidence of postoperative infections (e.g. epidural, subdural or subgaleal empyema). On the other hand, it is not known whether or not the application of TachoSil® on the dural suture may reduce CSF leakage.

ELIGIBILITY:
Inclusion Criteria:

* Neurosurgical indication for craniotomy and opening of dura to access cerebral structures/pathologies (discussed in the indication conference of board certified neurosurgeons at the University Hospital of Basel).
* The list of pathologies includes:

  * primary or secondary benign/malignant brain tumors
  * aneurysms
  * arterious-venous malformations
  * cavernomas
  * pituitary adenomas
  * temporal lobectomy (epilepsy surgery)
  * longterm posttraumatic revisions.

Exclusion Criteria:

* Presence of subdural empyema/abscess or any kind of infection affecting/infiltrating the dura mater
* Emergency for trauma
* Previous surgery on the same site
* Cases, where water-tight dural suture is not possible (intraoperative exclusion decision)
* Known hypersensitivity to TachoSil®
* Participation in another study
* Pregnancy
* Inability to read and understand the participant's information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2009-10; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Occurence of CSF pad or leakage needing any kind of intervention. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Mariani Luigi, Prof., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Derived] Hutter G, von Felten S, Sailer MH, Schulz M, Mariani L. Risk factors for postoperative CSF leakage after elective craniotomy and the efficacy of fleece-bound tissue sealing against dural suturing alone: a randomized controlled trial. J Neurosurg. 2014 Sep;121(3):735-44. doi: 10.3171/2014.6.JNS131917. Epub 2014 Jul 18. PMID 25036199